CLINICAL TRIAL: NCT01487291
Title: Prevalence of Clinical and Laboratory Markers of Hypofibrinolysis in Psychotic Patients
Status: Completed | Type: Observational
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Silvia Hoirisch Clapauch, MD, Responsible for the HFSE Thrombophilia Clinic, Universidade Federal do Rio de Janeiro
Other Study IDs: UFRiodJaneiro
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Insulin Resistance; Thrombophilia; Psychosis
Keywords: Thrombophilia tests; Hypofibrinolysis; Fibrinolysis
MeSH Terms: conditions — Insulin Resistance; Thrombophilia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Psychotic patients: Inpatients and outpatients followed at Instituto de Psiquiatria da Universidade Federal do Rio de Janeiro, Brazil

SUMMARY:
At the Thrombophilia Clinic of the Hospital Federal dos Servidores do Estado do Rio de Janeiro there is a high prevalence of acute psychotic episodes, which allows the investigators to raise the suspicion that the thrombotic tendency or hypofibrinolysis play a role in the onset of the disease. It is striking that most of these patients, after some time on anticoagulants, no longer need to take psychiatric medication.

DETAILED DESCRIPTION:
If the thrombotic tendency plays a significant role in the etiology of psychosis, one would expect to find ischemic brain injuries in neuroimaging studies, but it does not happen. Therefore, if there is a correlation between thrombotic tendency-hypofibrinolysis and psychosis it is likely to occur at the biochemical level, such as in neuronal transmission.

The investigators hypothesis is that mechanisms that inhibit tissue plasminogen activator (t-PA) and therefore promote hypofibrinolysis, are directly or indirectly involved in the genesis of psychosis, because t-PA participates in neuronal plasticity and low t-PA levels are related to dementia.

Hypofibrinolysis due to t-PA inhibition can be seen in:

* Insulin resistance, when the pancreas must produce large amounts of insulin and proinsulin by feedback. If pancreatic reserve is inadequate, the result is diabetes mellitus. If the response is adequate, proinsulin stimulates the production of PAI-1 (plasminogen activator inhibitor 1. PAI-1 inhibits the formation of plasmin, whose function is to dissolve fibrin which makes up the clot. Obesity, certain infections and inflammations potentiate insulin resistance.
* Antiphospholipid antibody syndrome.
* PAI-1 4G/5G or 4G/4G polymorphism.

Some hypofibrinolysis indicators are:

* severe dysmenorrhea, because strong uterine contractions are necessary to expel undissolved clots.
* PCOS because plasmin is required to activate some metalloproteinases involved in ovary remodelling.
* early pregnancy losses, as some metalloproteinases involved in placental angiogenesis are activated by plasmin,
* preeclampsia and eclampsia, as metalloproteinases that dissolve elastic fibers of the placental vessels, to create a low flow resistance, are activated by plasmin. Vascular endothelial growth factor (VEGF), a protein that restricts glomerular porosity, is also activated by plasmin,
* sudden death and heart attack before age 50 in first degree relatives.

On physical exam, acanthosis, high body mass index, and in women, hirsutism and acne are indirect indicators of insulin resistance. Livedo suggest antiphospholipid antibody syndrome.

This study intents to investigate the prevalence of hypofibrinolysis markers, such as PAI-1 4G/5G and 4G/4G, protein S deficiency, antiphospholipid antibodies and prothrombin G20210A, in psychotic patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder by the Semi-structured Interview MINI 5.0.

Exclusion Criteria:

* Inability to provide information.
* Use of illicit drugs.
* Infections such as cerebral toxoplasmosis in HIV seropositive or tertiary syphilis. Patients with "recurrent syphilis" will not be excluded, because false positive tests are common in antiphospholipid antibody syndrome.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Psychotic patients treated at IPUB-UFRJ, comprising patients with schizophrenia, schizoaffective disorders, bipolar disorders (mania or depressive episodes, provided that the patient has shown an acute psychotic episode in the last two years.
  Age-matched control group
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of hypofibrinolysis markers in psychotic patients | One year
  The investigators' hypothesis is that a high prevalence of hypofibrinolysis markers will be probably found in psychotic patients.

SECONDARY OUTCOMES:
Prevalence of Clinical and Laboratory Markers of Hypofibrinolysis in Patients who Need Electroconvulsive Therapy | 2013-2014
  The investigators are assessing clinical and laboratory markers of plasminogen activator imbalance in psychiatric patients who require electroconvulsive therapy, specifically patients with major depressive disorders and schizophrenia.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio E Nardi, MD, PhD, Study Chair — Universidade Federal do Rio de Janeiro, Brazil
Locations (1):
- Institudo de Psiquiatria da UFRJ, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Hoirisch-Clapauch S, Nardi AE. Multiple roles of tissue plasminogen activator in schizophrenia pathophysiology. Semin Thromb Hemost. 2013 Nov;39(8):950-4. doi: 10.1055/s-0033-1357505. Epub 2013 Oct 9. PMID 24108470
- [Background] Hoirisch-Clapauch S, Mezzasalma MA, Nardi AE. Pivotal role of tissue plasminogen activator in the mechanism of action of electroconvulsive therapy. J Psychopharmacol. 2014 Feb;28(2):99-105. doi: 10.1177/0269881113507639. Epub 2013 Oct 9. PMID 24113086
- [Result] Hoirisch-Clapauch S, Nardi AE. Markers of low activity of tissue plasminogen activator/plasmin are prevalent in schizophrenia patients. Schizophr Res. 2014 Oct;159(1):118-23. doi: 10.1016/j.schres.2014.08.011. Epub 2014 Sep 7. PMID 25205258